CLINICAL TRIAL: NCT01295710
Title: Phase 3 Study of US-ATG-F to Prevent Moderate to Severe Chronic GVHD in Adult Acute Myeloid Leukemia, Acute Lymphoid Leukemia, and Myelodysplastic Syndrome Patients After Allogeneic Stem Cell Transplantation From Unrelated Donors
Brief Title: Study of US-ATG-F to Prevent Chronic Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IV-ATG-SCT-01
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: GVHD; Adult Acute Myeloid Leukemia; Adult Acute Lymphoid Leukemia; Myelodysplastic Syndrome
Keywords: adult acute myeloid leukemia; adult acute lymphoid leukemia; adult myelodysplastic syndrome; allogenic stem cell transplantation; unrelated donor; GVHD; US-ATG-F (Anti-human-T-lymphocyte Immune Globulin, Rabbit)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- US-ATG-F (Active Comparator): 20 mg/kg body weight per day, diluted in 250 mL normal saline, IV infusion over 6-16 hours 3 days prior to transplantation
  Interventions: Biological: US-ATG-F
- Placebo (Placebo Comparator): 250 mL normal saline, IV infusion over 6-16 hours 3 days prior to transplantation
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: US-ATG-F — 20 mg/kg body weight per day, diluted in 250 mL normal saline, IV infusion over 6-16 hours 3 days prior to transplantation
  Other Names: Anti-human-T-lymphocyte Immune Globulin, Rabbit
  Arms: US-ATG-F
Biological: Placebo — 250 mL normal saline, IV infusion over 6-16 hours 3 days prior to transplantation
  Arms: Placebo

SUMMARY:
The study objective is to compare the efficacy and safety of US-ATG-F as a supplement to standard of care prophylaxis versus standard of care prophylaxis alone in moderate to severe chronic GVHD-free survival.

DETAILED DESCRIPTION:
This study is randomized, prospective, double-blind, placebo-controlled, phase 3 study evaluating the prevention of moderate to severe chronic GVHD in patients undergoing bone marrow or peripheral blood stem cell transplantation from matched, unrelated donors for acute leukemia and myelodysplastic syndrome during the first year after transplant.

Patients meeting all the inclusion and none of the exclusion criteria will be randomized (1:1). All patients will receive premedication and study drug 3 days prior to transplantation.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients designated to undergo allogeneic peripheral blood or bone marrow stem cell transplantation following the diagnosis of one of the primary diseases in early or intermediate disease status (i.e., acute myeloid leukemia, acute lymphoid leukemia, and myelodysplastic syndrome)
* Patients with an unrelated HLA-A,-B, -C and -DRBI matched donor
* Patients with a Karnofsky Performance Score ≥ 70%

Key Exclusion Criteria:

* Clinically significant concomitant diseases (i.e., cardiac, pulmonary, renal and CNS)
* Bacterial, viral, or fungal infections
* Known positive for Hepatitis B surfaces antigen, or Hepatitis C antibody, or who have been tested positive for HIV
* Patients with any concurrent malignancy. Cancer treated with curative intent < 5 years previously will not be allowed except for patients with resected basal cell carcinoma or treated cervical carcinoma in situ
* Known contraindications to the administration of rabbit immunoglobulin antibodies
* Hypersensitivity to methylprednisolone, tacrolimus, methotrexate or any excipients contains in these products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kuan, Study Director — Neovii Biotech
Locations (28):
- United States (26):
  - City of Hope, Duarte, California
  - Stanford University Medical Center, BMT, Stanford, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Abramson Cancer Center of the University at Perlman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Transplant Physician's Group, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - VA Puget Sound Healthcare System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria

REFERENCES:
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrollment number of 260 participants in the Protocol Section represents the number of patients who were randomized.
  The number of 254 participants who Started in the Participant Flow module represents the number of patients who were randomized and were treated.
Period: Overall Study
Arm/Group | US-ATG-F | Placebo
Started | 126 (Randomized and treated) | 128 (Randomized and treated)
Completed | 48 | 78
Not Completed | 78 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | US-ATG-F | Placebo | Total
Number analyzed (Participants) | 126 | 128 | 254
Age, Customized [Count of Participants; unit: Participants]
  18 years to ≤40 years | 42 | 43 | 85
  >40 years to 65 years | 84 | 85 | 169
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 49 | 115
  Male | 60 | 79 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 119 | 117 | 236
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 117 | 117 | 234
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 124 | 125 | 249
  Australia | 2 | 3 | 5
Disease [Count of Participants; unit: Participants]
  Acute lymphoid leukemia (ALL) | 23 | 34 | 57
  Myelodysplastic syndrome (MDS) | 19 | 14 | 33
  Acute myeloid leukemia (AML) | 83 | 80 | 163
  Biphenotypic AML/ALL | 1 | 0 | 1
Source of stem cells [Count of Participants; unit: Participants]
  Bone marrow | 22 | 27 | 49
  Peripheral blood | 95 | 101 | 196
  No stem cell transplantation | 9 | 0 | 9
Conditioning regimen [Count of Participants; unit: Participants]
  Cyclophosphamide & total body irradiation (CY-TBI) | 31 | 37 | 68
  Busulfan & cyclophosphamide (BU-CY) | 47 | 37 | 84
  Fludarabine & busulfan (FLU-BU) | 48 | 54 | 102
ALC at Study Day -3 Overall Study [Count of Participants; unit: Participants] — Participant's absolute lymphocyte count (ALC) prior to the start of study drug administration on Day -3, i.e. 3 days prior to stem cell transplantation
  Participants
    ALC ≤ 0.1 x 10^9 lymphocytes/L | 51 | 41 | 92
    ALC > 0.1 x 10^9 lymphocytes/L | 64 | 74 | 138
    Not tested | 11 | 13 | 24
ALC at Study Day -3 by Conditioning Regimen [Count of Participants; unit: Participants] — Participant's absolute lymphocyte count (ALC) prior to the start of study drug administration on Day -3, i.e. 3 days prior to stem cell transplantation. Participants are grouped based on administered conditioning regimen. Population: Analysis of patients who received a specific conditioning regimen
  Participants
    Regimen: CY-TBI: number analyzed (Participants) | 31 | 37 | 68
    Regimen: CY-TBI: ALC ≤ 0.1 x 10^9 lymphocytes/L | 22 | 24 | 46
    Regimen: CY-TBI: ALC > 0.1 x 10^9 lymphocytes/L | 7 | 11 | 18
    Regimen: CY-TBI: Not tested | 2 | 2 | 4
    Regimen: BU-CY: number analyzed (Participants) | 47 | 37 | 84
    Regimen: BU-CY: ALC ≤ 0.1 x 10^9 lymphocytes/L | 6 | 2 | 8
    Regimen: BU-CY: ALC > 0.1 x 10^9 lymphocytes/L | 39 | 31 | 70
    Regimen: BU-CY: Not tested | 2 | 4 | 6
    Regimen: FLU-BU: number analyzed (Participants) | 48 | 54 | 102
    Regimen: FLU-BU: ALC ≤ 0.1 x 10^9 lymphocytes/L | 23 | 15 | 38
    Regimen: FLU-BU: ALC > 0.1 x 10^9 lymphocytes/L | 18 | 32 | 50
    Regimen: FLU-BU: Not tested | 7 | 7 | 14
    Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91 | 186
    Regimens: BU-CY + FLU-BU: ALC ≤ 0.1 x 10^9 lymphocytes/L | 29 | 17 | 46
    Regimens: BU-CY + FLU-BU: ALC > 0.1 x 10^9 lymphocytes/L | 57 | 63 | 120
    Regimens: BU-CY + FLU-BU: Not tested | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Moderate to Severe Chronic GVHD According to 2005 NIH Criteria as Determined by the Independent Endpoint Committee or Death From Any Cause After Allogeneic Stem Cell Transplantation
Description: Participants with first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee or death from any cause after allogeneic stem cell transplantation, with a target of 124 total events of moderate or severe chronic GVHD, or death from any cause
Time Frame: Time from first study drug administration until the first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, or death from any cause, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 60 | 72

2. Secondary Outcome: Overall Survival
Description: Incidence of death from any cause
Time Frame: Time from first study drug administration until the occurrence of death from any cause, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 49 | 36

3. Secondary Outcome: Number of Participants With Chronic GVHD Mild to Severe
Description: Participants with the first occurrence of mild to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of mild to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 18 | 50

4. Secondary Outcome: Number of Participants With Chronic GVHD Moderate to Severe
Description: Participants with the first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 13 | 45

5. Secondary Outcome: Number of Participants With Chronic GVHD Severe
Description: Participants with the first occurrence of severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 3 | 16

6. Secondary Outcome: Number of Participants With Acute GVHD Grade I-IV
Description: Participants with the first occurrence of acute GVHD grade I-IV as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade I-IV as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 48 | 71

7. Secondary Outcome: Number of Participants With Acute GVHD Grade II-IV
Description: Participants with the first occurrence of acute GVHD grade II-IV as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade II-IV as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 28 | 53

8. Secondary Outcome: Number of Participants With Acute GVHD Grade III-IV
Description: Participants with the first occurrence of acute GVHD grade III-IV as determined by the Investigators, with death and re transplantation as competing risks
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade III-IV as determined by the Investigators, with death and re transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 8 | 17

9. Secondary Outcome: Number of Participants With Relapse
Description: Participants with relapse or disease recurrence, with death as competing risk
Time Frame: Time from first study drug administration until the occurrence of relapse, with death as competing risk, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 37 | 26

10. Secondary Outcome: Disease-free Survival
Description: Incidence of relapse or death
Time Frame: Time from first study drug administration until the occurrence of relapse or death, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 61 | 49

11. Secondary Outcome: Number of Participants With Transplant Related Mortality
Description: Participants with transplant related mortality
Time Frame: Time from first study drug administration until the occurrence of transplant related mortality, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 24 | 23

12. Secondary Outcome: Systemic Immunosuppressive Medication for Treatment of Moderate to Severe Chronic GVHD
Description: Participants who started on systemic immunosuppressive medicine for treatment of moderate to severe chronic GVHD as determined by the Investigator, with death and re-transplantation as competing risks
Time Frame: Time from first study drug administration until start of systemic immunosuppressive medicine for treatment of moderate to severe chronic GVHD as determined by the Investigator, with death and re-transplantation as competing risks, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 8 | 33

13. Post Hoc Outcome: Number of Participants With First Occurrence of Moderate or Severe Chronic GVHD According to 2005 NIH Criteria as Determined by Principal Investigator or Death From Any Cause After Allogeneic Stem Cell Transplantation
Description: Participants with first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators or death from any cause after allogeneic stem cell transplantation, with a target of 124 total events of moderate or severe chronic GVHD or death
Time Frame: Time from first study drug administration until the first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators or death from any cause, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 63 | 86

14. Post Hoc Outcome: Moderate to Severe Chronic GVHD-free, Relapse-free Survival (GRFS)
Description: Participants with moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death from any cause
Time Frame: Time from first study drug administration until the occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death from any cause, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 70 | 81

15. Post Hoc Outcome: Grade III-IV Acute GVHD-free, GRFS
Description: Participants with grade III-IV acute GVHD as determined by the Investigator, moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death from any cause
Time Frame: Time from first study drug administration until the occurrence of grade III-IV acute GVHD, moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death, assessed up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants | 72 | 85

16. Post Hoc Outcome: Number of Participants With First Occurrence of Moderate to Severe Chronic GVHD or Death From Any Cause by Conditioning Regimen
Description: Participants with first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee or death from any cause after allogeneic stem cell transplantation, with a target of 124 total events of moderate or severe chronic GVHD, or death from any cause. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 1
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 20 | 16
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 18 | 21
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 22 | 35
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 40 | 56

17. Post Hoc Outcome: Moderate to Severe Chronic GVHD-free, Relapse-free Survival (GRFS) by Conditioning Regimen
Description: Participants with moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death from any cause. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 14
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 23 | 20
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 21 | 22
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 26 | 39
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 47 | 61

18. Post Hoc Outcome: Grade III-IV Acute GVHD-free GRFS by Conditioning Regimen
Description: Participants with grade III-IV acute GVHD as determined by the Investigator, moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Independent Endpoint Committee, relapse or death from any cause. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 15
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 23 | 21
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 23 | 22
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 26 | 42
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 49 | 64

19. Post Hoc Outcome: Overall Survival by Conditioning Regimen
Description: Incidence of death from any cause. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the occurrence of death from any cause, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 17 | 8
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 12 | 8
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 20 | 20
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 32 | 28

20. Post Hoc Outcome: Chronic GVHD Mild to Severe by Conditioning Regimen
Description: Participants with the first occurrence of mild to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 3
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 7 | 16
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 6 | 14
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 5 | 20
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 11 | 34

21. Post Hoc Outcome: Chronic GVHD Moderate to Severe by Conditioning Regimen
Description: Participants with the first occurrence of moderate to severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 4
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 5 | 13
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 6 | 13
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 2 | 19
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 8 | 32

22. Post Hoc Outcome: Chronic GVHD Severe by Conditioning Regimen
Description: Participants with the first occurrence of severe chronic GVHD according to 2005 NIH criteria as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 5
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 1 | 5
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 1 | 4
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 1 | 7
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 2 | 11

23. Post Hoc Outcome: Acute GVHD Grade I-IV by Conditioning Regimen
Description: Participants with the first occurrence of acute GVHD grade I-IV as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade I-IV, with death and re transplantation as competing risks, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 13 | 18
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 19 | 23
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 16 | 30
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 35 | 53

24. Post Hoc Outcome: Acute GVHD Grade II-IV by Conditioning Regimen
Description: Participants with the first occurrence of acute GVHD grade II-IV as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade II-IV, with death and re transplantation as competing risks, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 8 | 14
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 12 | 17
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 8 | 22
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 20 | 39

25. Post Hoc Outcome: Acute GVHD Grade III-IV by Conditioning Regimen
Description: Participants with the first occurrence of acute GVHD grade III-IV as determined by the Investigators, with death and re transplantation as competing risks. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the first occurrence of acute GVHD grade III-IV, with death and re transplantation as competing risks, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 3 | 2
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 4 | 5
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 1 | 10
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 5 | 15

26. Post Hoc Outcome: Relapse by Conditioning Regimen
Description: Participants with relapse or disease recurrence, with death as competing risk. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the occurrence of relapse with death as competing risk, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 11 | 6
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 8 | 7
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 18 | 13
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 26 | 20

27. Post Hoc Outcome: Disease-free Survival by Conditioning Regimen
Description: Incidence of relapse or death. Analysis was conducted by conditioning regimen.
Time Frame: Time from first study drug administration until the occurrence of relapse or death, assessed up to 48 months
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 21 | 13
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 15 | 11
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 25 | 25
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 40 | 36

28. Post Hoc Outcome: Transplant-related Mortality by Conditioning Regimen
Description: Participants with transplant related mortality. Analysis was conducted by conditioning regimen.
Time Frame: as for outcome 11
Population: Analysis of patients who received a specific conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | US-ATG-F | Placebo
Number analyzed (Participants) | 126 | 128
Participants
  Regimen: CY-TBI: number analyzed (Participants) | 31 | 37
  Regimen: CY-TBI | 10 | 7
  Regimen: BU-CY: number analyzed (Participants) | 47 | 37
  Regimen: BU-CY | 7 | 4
  Regimen: FLU-BU: number analyzed (Participants) | 48 | 54
  Regimen: FLU-BU | 7 | 12
  Regimens: BU-CY + FLU-BU: number analyzed (Participants) | 95 | 91
  Regimens: BU-CY + FLU-BU | 14 | 16

ADVERSE EVENTS:
Arm/Group | US-ATG-F | Placebo
Serious Adverse Events (participants affected / at risk) | 98/126 | 90/128
Other Adverse Events (participants affected / at risk) | 125/126 | 126/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | US-ATG-F (N=126) | Placebo (N=128)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11) | 6 (6)
Haemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 6 (6) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 7 (8)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastropleural fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10) | 7 (7)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8) | 8 (8)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (1)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 4 (4) | 5 (5)
Multi-organ failure (General disorders) | 5 (5) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 13 (14) | 15 (20)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 6 (6) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Acute graft versus host disease in intestine (Immune system disorders) | 1 (2) | 3 (3)
Chronic graft versus host disease (Immune system disorders) | 0 (0) | 3 (3)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 0 (0)
Engraftment syndrome (Immune system disorders) | 0 (0) | 2 (2)
Graft versus host disease (Immune system disorders) | 2 (2) | 5 (5)
Graft versus host disease in lung (Immune system disorders) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (4) | 4 (4)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4) | 4 (4)
Clostridial infection (Infections and infestations) | 2 (2) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (3)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis viral (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus chorioretinitis (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (2)
Cytomegalovirus infection (Infections and infestations) | 4 (4) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 4 (4)
Encephalitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis herpes (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 2 (3) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 3 (4) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 2 (2) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal abscess central nervous system (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Fusobacterium infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9) | 14 (22)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 4 (4)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Pyothorax (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (6) | 13 (13)
Septic shock (Infections and infestations) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 5 (5) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Systemic mycosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral haemorrhagic cystitis (Infections and infestations) | 3 (4) | 0 (0)
Zygomycosis (Infections and infestations) | 1 (1) | 0 (0)
Delayed engraftment (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 3 (3)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0)
Legionella test positive (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Polyomavirus test positive (Investigations) | 1 (1) | 1 (1)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0)
Respiratory syncytial virus test positive (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Acute myeloid leukemia, recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 5 (5)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 5 (6)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 4 (4)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | US-ATG-F (N=126) | Placebo (N=128)
Nausea (Gastrointestinal disorders) | 54 (63) | 47 (56)
Vomiting (Gastrointestinal disorders) | 38 (43) | 24 (27)
Diarrhoea (Gastrointestinal disorders) | 36 (45) | 22 (28)
Stomatitis (Gastrointestinal disorders) | 25 (26) | 26 (26)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 11 (11)
Constipation (Gastrointestinal disorders) | 2 (2) | 8 (8)
Mucosal inflammation (General disorders) | 41 (44) | 41 (47)
Pyrexia (General disorders) | 57 (71) | 1 (2)
Fatigue (General disorders) | 33 (36) | 34 (34)
Chills (General disorders) | 50 (54) | 7 (7)
Oedema peripheral (General disorders) | 11 (11) | 3 (3)
Pain (General disorders) | 10 (10) | 2 (6)
Cytomegalovirus infection (Infections and infestations) | 12 (16) | 18 (20)
Cytomegalovirus viraemia (Infections and infestations) | 13 (19) | 10 (12)
Epstein-Barr virus infection (Infections and infestations) | 14 (16) | 6 (7)
Clostridial infection (Infections and infestations) | 5 (7) | 7 (8)
Clostridium difficile colitis (Infections and infestations) | 11 (13) | 2 (3)
Staphylococcal bacteraemia (Infections and infestations) | 9 (13) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (9) | 3 (3)
Epstein-Barr viraemia (Infections and infestations) | 8 (8) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 34 (44) | 47 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (42) | 12 (29)
Anaemia (Blood and lymphatic system disorders) | 14 (27) | 11 (21)
Neutropenia (Blood and lymphatic system disorders) | 12 (22) | 8 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
White blood cell count decreased (Investigations) | 9 (15) | 5 (9)
Blood bilirubin increased (Investigations) | 9 (14) | 2 (3)
Epstein-Barr virus test positive (Investigations) | 7 (7) | 1 (3)
Headache (Nervous system disorders) | 38 (44) | 19 (22)
Dizziness (Nervous system disorders) | 8 (10) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 31 (35) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Hypotension (Vascular disorders) | 32 (36) | 6 (7)
Hypertension (Vascular disorders) | 16 (17) | 6 (6)
Flushing (Vascular disorders) | 9 (9) | 2 (2)
Tachycardia (Cardiac disorders) | 23 (24) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 19 (19) | 5 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 13 (13) | 6 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 16 (30) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No